CLINICAL TRIAL: NCT03269838
Title: Correlation of QT Dispersion With Myocardial Perfusion in Patients With ST Elevation Myocardial Infarction Treated by Primary Per Cutaneous Coronary Intervention
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, MS Roshdy, Principal Investigator, Assiut University
Other Study IDs: 17100310
Record Dates: First submitted 2017-08-27; First posted 2017-09-01 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: ST Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Electrocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ECG — Primary Percutaneous coronary intervention
  Other Names: Primary Percutaneous coronary intervention

SUMMARY:
To correlate QT dispersion on 12-lead surface ECG with myocardial reperfusion evaluated by myocardial blush grade and Thrombolysis in myocardial infarction (TIMI) flow grades in patients with ST elevation myocardial infarction treated by Primary Per cutaneous coronary intervention

DETAILED DESCRIPTION:
Worldwide, coronary artery disease (CAD) is the most frequent cause of death. Over seven million people every year die from CAD, accounting for 12.8% of all deaths. Every sixth man and every seventh woman in Europe die from myocardial infarction. The in-hospital mortality of STEMI patients in the national registries of the European society of cardiology (ESC) countries varies between 6% and 14%.

ST elevation myocardial infarction (STEMI) generally results from intraluminal thrombus formation and occlusion of a ruptured or an unstable plaque .

The main goal of therapy in STEMI is to restore microvascular flow and sustain the myocardial perfusion .

Reperfusion therapy for acute myocardial infarction (AMI) is aimed at achieving prompt restoration of myocardial perfusion to maximize preservation of the electrical and mechanical integrity of the jeopardized myocardium. Percutaneous coronary intervention (PCI) has increased the rate of successful recanalization of infarct-related arteries (IRAs) to >90% .

A variety of markers including ECG and coronary angiography have been utilized to assess myocardial reperfusion .

The prolongation of QRS duration,evaluated by a standard 12-lead ECG, is a marker of ventricular dysfunction and has been associated with a poor prognosis in STEMI .

QT-interval parameters are potentially proposed as available non-invasive markers for assessing the ventricular homogeneity as well as for predicting electrical instability ,QT interval (QTI) is defined as the longest interval from the beginning of the QRS complex to the end of the T-wave; QT dispersion (QTd) is defined as the difference between the longest and shortest QTI, and reflects electrical activity of the ventricles . .

The prolongation of the latter parameter is a main predictor for fatal arrhythmia in patients with myocardial infarction (MI) .

The measurement of QTI and QTd parameters are dependent on heart rate and can be corrected by the QT correction formulas, which are termed the corrected QTI (QTc) and QTd (QTcd) .

Myocardial blush grade (MBG) is validated measurement of myocardial perfusion . The MBG is used to assess the washout of myocardial blush during angiography. Grade 0 is defined as the failure of the contrast to enter the microvasculature. In grade 1 cases, contrast enters slowly, but fails to exit the microvasculature. Grade 2 defines delayed entry and exit from the microvasculature. Finally, grade 3 indicates normal entry and exit from the microvasculature .

ECG is a necessary, simple, rapid and non invasive tool for the diagnosis of myocardial infarction and evaluation of myocardial reperfusion that still to be investigated . QT dispersion is a crude and approximate measure of a general abnormality of repolarization; it reflects inhomogeneity of ventricular repolarization . This measurement is an attempt to distinguish between myocardium that is homogeneous from myocardium that displays inhomogeneity, which is accompanied by increased dispersion of the ventricular recovery times and prolongation of repolarization

ELIGIBILITY:
Inclusion Criteria:

* Patients will be enrolled in this study if they fulfilled the criteria of acute ST elevation myocardial infarction eligible to be treated with primary Percutaneous coronary intervention

Exclusion Criteria:

1. Non-ST elevation myocardial infarction, prior history of myocardial infarction or surgical revascularization,
2. Electrolyte disturbance.
3. history of medications that may affect QT (anti-arrhythmic, anti-psychotic, and anti-depressant drugs),
4. patients with cardiogenic shock or needing IABP.
5. patients with previous CABG.
6. Patients with implantable devices and pacemakers.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: This cross sectional observational study will include patients with acute STEMI of different ages from cardiology department, Assiut University Hospital who will undergo primary percutaneous coronary intervention (PCI).
Sampling Method: Probability Sample
Enrollment: 235 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Correlation of QT dispersion on 12-lead surface ECG with myocardial reperfusion | 1 year
  Use 12 lead ECG to calculate QT interval and QT dispersion comparing ECG before and after myocardial reperfusion.
Evaluation of myocardial perfusion by coronary angiography by assessing 2 parameters TIMI flow and myocardial blush grade | 1 year
  Use coronary angiography to detect myocardial blush grade and TIMI flow to assess myocardial reperfusion

CONTACTS AND LOCATIONS:
Overall Officials: Hatem Helmy, Study Chair — assistant professor; Hosam Hasan, Study Chair — professor
Locations (1):
- Assiut university, Asyut, Egypt

REFERENCES:
- [Background] Karahan Z, Yaylak B, Ugurlu M, Kaya I, Ucaman B, Ozturk O. QRS duration: a novel marker of microvascular reperfusion as assessed by myocardial blush grade in ST elevation myocardial infarction patients undergoing a primary percutaneous intervention. Coron Artery Dis. 2015 Nov;26(7):583-6. doi: 10.1097/MCA.0000000000000285. PMID 26166018